CLINICAL TRIAL: NCT02134080
Title: FAAH Inhibitor Trial for Adults With Tourette Syndrome
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: no more funding available
Sponsor: Yale University (Other)
Collaborators: Tourette Association of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1403013669
Record Dates: First submitted 2014-05-06; First posted 2014-05-08 (Estimated); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; FAAH-Inhibitor; Tics; Tic Disorders
MeSH Terms: conditions — Tourette Syndrome; Tics; Tic Disorders | interventions — N-pyridazin-3-yl-4-(3-((5-(trifluoromethyl)pyridin-2-yl)oxy)benzylidene)piperidine-1-carboxamide; fatty-acid amide hydrolase; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- PF-04457845 (Active Comparator): PF-04457845 will be administered orally at 4mg daily for four weeks.
  Interventions: Drug: PF-04457845
- Placebo (Placebo Comparator): Placebo (sugar pill) will be administered orally at 4mg daily for four weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04457845 — PF-04457845 will be administered orally at 4mg daily for four weeks.
  Other Names: fatty acid amide hydrolase (FAAH) inhibitor
  Arms: PF-04457845
Drug: Placebo — Placebo will be administered orally at 4mg daily for four weeks.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this trial is to examine the safety, tolerability and feasibility in the use of a FAAH inhibitor for the treatment of adults with Tourette syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Adult between 18-60 years of age
* Meet DSM IV criteria for the diagnosis of Tourette's syndrome
* Significant current tic symptoms: YGTSS total tic score greater than or equal to 22 at baseline
* On stable psychiatric medication regimen for a minimum of 4 weeks prior to beginning the trial.
* Accepted method of birth control

Exclusion Criteria:

* Comorbid bipolar disorder, psychotic disorder, substance use disorder, developmental disorder or intellectual disability (IQ<70).
* Current use of medications that have significant effects on the cannabinoid or dopamine systems. Subjects will be specifically excluded for recent use (within last 8 weeks) of antipsychotic medications, dopamine agonists or psychostimulants.
* Recent change (less than 4 weeks) in other medications that have potential effects on tic severity (such as alpha-2 agonists (guanfacine, clonidine or prazosin), SSRIs, clomipramine, naltrexone, lithium, anxiolytics, topiramate, baclofen etc.). Medication change is defined to include dose changes or medication discontinuation.
* Recent change in behavioral treatment for Tourette syndrome or comorbid conditions (i.e. OCD) within the last 4 weeks or initiation of behavioral therapy for tics within the last 12 weeks.
* Positive pregnancy test or drug screening test
* History of cannabis dependence
* Significant Medical Comorbidity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Improvement in Tic Severity | Evaluated each time subject seen over approximately 12 weeks
  Yale Global Tic Severity Scale (Total Tic Score)

SECONDARY OUTCOMES:
Improvement of Premonitory Urges | Evaluated each time subject seen over approximately 12 Weeks
  Premonitory Urge for Tics Scale (PUTS)
Improvement in Obsessive Compulsive Disorder (OCD) Severity | Evaluated every two weeks over the course of approximately 12 weeks
  Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)
Self-Report of Tic Severity | Evaluated each time subject seen over approximately 12 weeks
  Tourette Syndrome Symptom List (TSSL)
Video-Tape Ratings of Tic Severity | Evaluated every two weeks over the course of approximately 12 weeks
  Modified Rush Video Rating Scale
ADHD Severity | Evaluated every two weeks over the course of approximately 12 weeks
  Connors Adult Attention Deficit Hyperactivity Rating Scale
Depression Severity | Evaluated every two weeks over the course of approximately 12 weeks
  Hamilton Rating Scale for Depression
Anxiety Severity | Evaluated every two weeks over the course of approximately 12 weeks
  Hamilton Rating Scale for Anxiety
Overall improvement | Evaluated each time subject seen over approximately 12 Weeks
  Clinical Global Improvement Scale
Number of Adverse Events | Evaluated each time subject seen over approximately 12 Weeks
  Adverse Events Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael H. Bloch, MD, MS, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States